CLINICAL TRIAL: NCT02902224
Title: Glucose and Fructose Stimulated Brain Activity in Obese Subjects Before and After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: fMRI BARI
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Exploratory Behavior
MeSH Terms: conditions — Exploratory Behavior | interventions — Glucose; Fructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PLACEBO (Placebo Comparator): Single intragastric instillation of 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Tap water
- GLUCOSE (Active Comparator): Single intragastric instillation of 75g Glucose in 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Glucose
- FRUCTOSE (Active Comparator): Single intragastric instillation of 25g Fructose in 300ml tap water via nasogastric tube
  Interventions: Dietary Supplement: Fructose

INTERVENTIONS:
Dietary Supplement: Tap water — 300ml tap water via nasogastric tube
  Arms: PLACEBO
Dietary Supplement: Glucose — 300ml tap water with 75g glucose via nasogastric tube
  Arms: GLUCOSE
Dietary Supplement: Fructose — 300ml tap water with 25g fructose via nasogastric tube
  Arms: FRUCTOSE

SUMMARY:
The objective is to investigate neuro-anatomical correlates of the regulation of energy intake by means of functional MRI before and after bariatric surgery. Administration of glucose as well as fructose is followed by functional brain MRI, and findings are correlated with serum glucagon-like peptide 1 (GLP-1) levels as an endogenous satiety signal in obese humans.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* morbidly obese patients
* scheduled for bariatric surgery

Exclusion Criteria:

* Diabetes mellitus
* cardiovascular disease
* neurologic or psychiatric disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) in healthy, obese volunteers while they performed a working memory task: changes in cerebral blood flow | changes from baseline to one hour after treatment

SECONDARY OUTCOMES:
Changes in plasma glucose | Changes from baseline to one hour after treatment
Changes in plasma insulin | Changes from baseline to one hour after treatment
Changes in Plasma GLP-1 | Changes from baseline to one hour after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof, Study Chair — University of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided